CLINICAL TRIAL: NCT04884256
Title: A Phase 2 Multicenter, Randomized, Vehicle-Controlled Study to Evaluate the Safety and Efficacy of CBT-004 Ophthalmic Emulsion in Patients With Vascularized Pinguecula
Brief Title: Safety and Efficacy Study of CBT-004 in Patients With Vascularized Pinguecula
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cloudbreak Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CBT-CS103
Record Dates: First submitted 2021-05-05; First posted 2021-05-12 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-02

CONDITIONS: Pinguecula
MeSH Terms: conditions — Pinguecula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CBT-004 (Placebo Comparator)
  Interventions: Drug: CBT-004
- 0.05% CBT-004 (Experimental)
  Interventions: Drug: CBT-004
- 0.075% CBT-004 (Experimental)
  Interventions: Drug: CBT-004

INTERVENTIONS:
Drug: CBT-004 — Dose response study

SUMMARY:
STUDY DESIGN:

Structure:

Multicenter, randomized, double-masked, vehicle-controlled, parallel-group study.

Duration of Treatment:

4 weeks of study treatment with 4 weeks follow-up observations.

Control:

Vehicle for CBT-004 (hereafter referred to as Vehicle).

Masking:

Subjects, Investigators, Study Monitors and the Independent Image Reading Center are all masked to the study medications.

Dosage/Dose regimen:

One drop of the assigned study medication will be administered in the study eye TID for 4 weeks. The study eye is defined as the qualified eye (i.e., the eye meeting the inclusion criterion for vascularized pinguecula). If both eyes are qualified, then the eye with the more severe vascularity grade at Visit 1 will be the study eye.

ELIGIBILITY:
Inclusion Criteria:

* Pinguecula with a vascularity grade ≥ 3 on a 5-point (0-4) scale.
* Ocular bothersome questionnaire score ≥ 2 on a 5-point (0-4) scale.
* ≥ 18 years of age.
* Able to provide written informed consent and comply with study assessments for the full duration of the study.

Exclusion Criteria:

* Uncontrolled systemic disease, in the opinion of the investigator.
* Active ocular disease other than pinguecula that may confound the study data, including but not limited to severe dry eye disease, pterygium, uncontrolled blepharitis, anterior membrane dystrophy, Salzmann's, glaucoma, or active ocular infection.
* History of ocular herpes disease, iritis/uveitis, in either eye.
* Any ocular surgical procedure within the last 3 months or anticipated ocular surgery during the study, in either eye.
* Anticipated wearing of contact lenses during any portion of the study. Patients, who wear soft contact lenses should discontinue wearing them at least 7 days prior to Day 1 visit. Patients wearing rigid gas permeable or hard contact lenses should discontinue wearing them at least 3 weeks prior to Day 1 visit.
* Female patients who are pregnant, nursing, or planning a pregnancy during the study.
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days prior to entry into this study.
* History of myocardial infarction or stroke.
* Any condition or situation which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study.
* Known allergy or sensitivity to the study medication(s) or its components.
* Current or anticipated use of topical ophthalmic medications in the study eye. Patients must have discontinued use of ophthalmic medications in the study eye for at least 2 weeks (4 weeks for Restasis® or Xiidra®) prior to Day 1 visit. Artificial tears are allowed in the study eye until 7 days prior to Visit 1 and should not be used during the treatment phase of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in conjunctival hyperemia grade at Day 28 (Week 4). | 1 month

SECONDARY OUTCOMES:
Change from Baseline conjunctival hyperemia digital image grade at Days 7 (Week 1) and 56 (Week 8). | 2 month

CONTACTS AND LOCATIONS:
Locations (1):
- Global Research Management, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Undecided